CLINICAL TRIAL: NCT03002636
Title: Safety and Risk Assessment of Obese Parturient Underwent Cesarean Section(CS) Delivery Under General Anesthesia or Intraspinal Anesthesia
Brief Title: Safety and Risk Assessment of Obese Parturient Underwent Cesarean Section(CS) Delivery Under Different Anesthesia Ways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Zeyong Yang, International Peace Maternity and Child Health Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IPMCH-anes
Record Dates: First submitted 2016-12-07; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Cesarean Section
Keywords: Obesity; Anesthesia Complications; Body Mass Index (BMI)
MeSH Terms: conditions — Obesity | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Morbid Obesity group (Experimental): Morbid Obesity group(n=300)
  Interventions: Procedure: anesthesia
- severe Obesity group (Experimental): severe Obesity group (n=300)
  Interventions: Procedure: anesthesia
- non-Obesity group (Other): non-Obesity group(n=300)
  Interventions: Procedure: anesthesia

INTERVENTIONS:
Procedure: anesthesia — Anesthesia : (1) General Anesthesia (GA)(2) Epidural Anesthesia (EA) (3) Combined Spinal-Epidural Anesthesia (CSEA)

SUMMARY:
900 parturient who underwent CS under general anesthesia(GA) , intraspinal anesthesia included epidural anesthesia(EA) and combined spinal-epidural anesthesia(CSEA), which were divided into 3 groups: Morbid Obesity group (n=300) with body mass index (BMI) >40 kg/m2 , severe Obesity group (n=300) with 30 kg/m2≤BMI ≤40 kg/m2 and non-Obesity group(n=300) with BMI<30 kg/m2. Findings Between January 1, 2013 and September 30, 2016, a total of 1000 women met inclusion criteria and 900 women received allocated intervention. All patients were divided into three groups: Morbid Obesity group(n=300), Severe Obesity group(n=300) and non-Obesity group(n=300) according to body mass index (BMI) >40 kg/m2, 30 kg/m2≤BMI ≤40 kg/m2 and BMI<30 kg/m2.900 patients completed the protocol and related data were analysed.

DETAILED DESCRIPTION:
900 parturient who underwent CS under general anesthesia(GA) , intraspinal anesthesia included epidural anesthesia(EA) and combined spinal-epidural anesthesia(CSEA), which were divided into 3 groups

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA Physical Status gradeΙΙ～ΙΙΙ.

Exclusion Criteria:

* scoliosis, congenital heart disease, lung, liver, kidney diseases or increased intracranial pressure (ICP)

Ages: 24 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patients numbers of obese parturient complications | 2 years
  Patients numbers of emergency, fetal macrosomia, gestational diabetes mellitus (GMD), CS history, fetal distress, elderly parturient women(≥35 years), prenatal fever, arrhythmias, abnormalities of the heart, hypertension(pre-eclampsia), multiple pregnancy, precious child, amniotic fluid abnormality, amout of bleeding, neonate Apgar's Score(1min), Apgar's Score(5min), and patients numbers of EA, GA, PACU (Postanesthesia Care Unit ) and ICU (Intensive Care Unit) for duration of hospital stay and anesthesia puncture times with 5>n≥3 and n≥5 in three groups included non-Obesity group, severe Obesity group and Morbid Obesity group were also recorded. In addition, we also recorded puncture patients numbers in sitting position for all groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Gao, MD, Study Director — Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An X, Zhao Y, Zhang Y, Yang Q, Wang Y, Cheng W, Yang Z. Risk assessment of morbidly obese parturient in cesarean section delivery: A prospective, cohort, single-center study. Medicine (Baltimore). 2017 Oct;96(42):e8265. doi: 10.1097/MD.0000000000008265. PMID 29049219